CLINICAL TRIAL: NCT03761355
Title: Mindfulness and Executive Functions for Prediction of Non-technical Skills of Students in High-fidelity Medical Simulations in Pediatric Emergency Cases
Brief Title: Mindfulness and Executive Functions for Prediction of Non-technical Skills of Students in Pediatric Medical Simulations
Acronym: MindExSim
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Other Study IDs: N/ST/ZB/18/002/1206
Record Dates: First submitted 2018-11-19; First posted 2018-12-03 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Mindfulness
Keywords: mindfulness; executive functions; medical simulation; medical students; pediatrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- medical student of 6th Year: Students of medical faculty of 6th Year in Medical University of Bialystok, Poland.

SUMMARY:
Medical simulation is a technique that creates a situation or environment to allow persons to experience a representation of a real event for the purpose of practice, learning, evaluation, testing or to gain understanding of systems or human actions Non-technical skills in pediatric simulation are the skills of communication, leadership, teamwork, situational awareness, decision-making, resource management, safe practice, adverse event minimization, and professionalism, also known as teamwork skills. Mindfulness is the self-regulation of attention with an attitude of curiosity, openness and acceptance. Executive functions include a collection of interrelated functions that are responsible for purposeful, goal-directed, problem-solving behavior. In this project, the investigators aim to check whether features of mindfulness and executive functions can be used to predict teamwork skills of medical students during repeated high-fidelity simulations in emergency pediatric care.

The project will include simulation center in Bialystok, Poland. The investigators will conduct this project over a time of 2 years. Team project is made up of 5 persons, including psychologist, simulation instructors and pediatricians. Participants will be students of medical faculty in medical university. The investigators expect to include at least 340 students in the study which will result in 180 assessed as main or second leaders in repeated simulations. Team project will assess the students during high-fidelity pediatric emergency simulations.

Methods of assessment of medical students during pediatric emergency simulations: features of mindfulness (Mindful Attention Awareness Scale), assessment of executive functions (The Behavior Rating Inventory of Executive Functions - Adult), non-technical skills (Ottawa Crisis Resource Management scale & checklist), technical skills (checklists) and stress. The researchers first will examine association between mindfulness or executive functions and demographic variables. And finally team project will assess the possibility of prediction of non-technical performance level during medical simulations with the use of mindfulness and executive functions assessment.

In general the investigators anticipate that the results of the study will lead to the better understanding of mechanisms that influence non-technical skills in medical students during pediatric emergency cases.

DETAILED DESCRIPTION:
Research Project Objectives / Research Hypothesis High-fidelity simulation is an effective tool in creating psychological reality of pediatric emergency care. Non-technical skills play a pivotal role in management of life-threatening cases in children. Mindfulness is the self-regulation of attention with an attitude of curiosity, openness and acceptance. It is possible that mindfulness could enhance medical students' capacity for focused attention and concentration by increasing present moment awareness. On the other hand executive functions include a collection of interrelated functions that are responsible for purposeful, goal-directed, problem-solving behavior. It is likely that mindfulness and executive functions and their relationship are important players in emergency cases. Repeated simulations could be a crucial tool for stress management and improving skills in high-fidelity scenarios. In this project, the investigators aim to define whether features of mindfulness and executive functions can be used to predict non-technical skills of medical students during repeated high-fidelity simulations in emergency pediatric care. The researchers hypothesize that: 1) being mindful improves the performance during simulation 2) better executive functions result in better non-technical skills of medical student 3) repeated simulations will reduce stress and influence performance during scenarios 4) there are some potential correlations between executive functions and mindfulness 5) it is possible to predict non-technical performance with the assessment of mindfulness and executive functions of students during pediatric emergency cases.

Research project methodology This is a multi-center, investigator-initiated prospective study. The project will include simulation center in Poland (Medical University in Białystok). The researchers will conduct this project over a time of 2 years. Team project is made up of 5 persons, including psychologist, simulation instructors and pediatricians. Participants will be students of medical faculty in medical university. Methods: First, to increase the awareness of scientific community of the area of interest, the scientists will prepare and publish the review of the current literature in the field of mindfulness, executive functions and emergency medicine. Then, the researchers will adapt six high-fidelity scenarios in the field of pediatric emergency for the requirements of the project. The team project expect to include at least 340 students in the study which will result in 180 assessed as main or second leaders in repeated simulations. For the accomplishment of the aims of this study researchers will need: high-fidelity simulation rooms = emergency rooms with full medical equipment, high-fidelity simulators, audio-video systems for recording and playing scenarios, ECG Holters, debriefing rooms, computers and software. All above mentioned equipment is available in simulation centers and the investigators have the professional staff experienced in high-fidelity simulation and assessment of non-technical skills in medical students. Demographic features will be assessed in all participants: age, sex, year of medical faculty, medical school. The history of previous high-fidelity simulations in participating students will be collected. Methods of assessment of medical students during pediatric emergency simulations: features of mindfulness (Mindful Attention Awareness Scale), assessment of executive functions (The Behavior Rating Inventory of Executive Functions - Adult), non-technical skills (Ottawa Crisis Resource Management scale & checklist), technical skills (checklists) and stress (heart rate, heart rate variability with Holter ECG, blood pressure, Stress-O-Meter and the State-Trait-Anxiety Inventory). Data analysis strategy: The study team will first examine association between mindfulness or executive functions and demographic variables (gender, age, university). Then the researchers are going to construct the regression model to explain the variability of features included in Ottawa scale. And finally the study team will assess the possibility of prediction of non-technical performance level during medical simulations with the use of mindfulness and executive functions assessment.

Expected impact of the research project on the development of science To date more than 150 students were enrolled for the preliminary research. The preliminary results showed that: in the first simulation the students' non-technical performance is weak, one of the main problems in non-technical skills is the fixation error and it is more frequent in simulations with two cases at one time, in the repeated simulations non-technical skills are improving, there is a growing interest in mindfulness training among medical students, technical skills depend of theoretical introduction and students' preparation for the classes, concerning stress the statistically significant increase in heart rate but not blood pressure in students after each simulation was observed . These data clearly show that the proposed study concept is a promising line of basic investigation with solid potential for defining a predictive link between mindfulness, executive function and non-technical skills of medical students during pediatric emergency simulations. In general the investigators anticipate that the results of the present study will lead to the better understanding of mechanisms that influence non-technical skills in medical students during pediatric emergency cases. In the future this research will be used for an overall improvement in team performance at emergency events, which will ultimately translate into a subsequent reduction in the rate of errors and adverse events in medicine. The team leaders also hope that an increased awareness of non-technical skills in the emergency setting among medical students will have an indirect beneficial effect on those skills in the day-to-day setting.

The scientific results of the project will include: review manuscript and at least two original manuscripts, all published in Journals with Impact Factor ≥ 3, presentations on two international meetings in Europe.

ELIGIBILITY:
Inclusion Criteria:

* student of 6th Year of medical faculty
* informed consent

Exclusion Criteria:

* pregnancy

Ages: 23 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students of medical faculty (6th year) at the Medical University of Bialystok
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Non-technical skills - Ottawa scale | 12 months
  We have chosen Ottawa Ottawa Crisis Resource Management Global Rating Scale to evaluate performance during our simulations. The following criteria will be evaluated: leadership skills (stays calm and in control during crisis, prompt and firm decision-making, maintains global perspective - "big picture"), situational awareness (avoids fixation error, reassesses and re-evaluates situation constantly, anticipates likely events), communication skills (communicates clearly and concisely, uses directed verbal /non-verbal communication, listens to team input), problem solving (organized and efficient problem solving approach, quick in implementation, considers alternatives during crisis), resource utilization (calls for help appropriately, utilizes resources at hand appropriately, prioritizes tasks appropriately). Each category is measured on a seven-point anchored ordinal scale with descriptive anchors. The higher values represent a better outcome.

SECONDARY OUTCOMES:
Technical skills | 12 months
  Technical skills of medical students during high-fidelity simulations. We designed and validated a scale for assessment technical skills in each scenarios. An example is presented below. The higher values represent a better outcome.
  An example of newly developed technical skills checklist for the use in this project - topic - "Ketoacidosis"
  Action:
  * History - including polydypsia (1 point), polyuria (1 point), weight loss (1 point)
  * Physical examination: breathing, pulse, blood pressure, saturation, heart and lung auscultation, abdomen, dehydration
  * Treatment:
    * Hydratation 0.9%NaCl i.v.1000ml / first hour (1 point)
    * Insulin (rapid acting, 0.1Units/kg) iv (1 point)
    * Potassium (15%KCl 10-20mmol) (1 point)
    * No addition of Natrium carbonicum (1 point)

CONTACTS AND LOCATIONS:
Overall Officials: Wlodzimierz Luczynski, Prof, Study Chair — Medical University of Bialystok
Locations (1):
- Medical University of Bialystok, Bialystok, Podlaskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eppich WJ, Brannen M, Hunt EA. Team training: implications for emergency and critical care pediatrics. Curr Opin Pediatr. 2008 Jun;20(3):255-60. doi: 10.1097/MOP.0b013e3282ffb3f3. PMID 18475092
- [Background] Jirativanont T, Raksamani K, Aroonpruksakul N, Apidechakul P, Suraseranivongse S. Validity evidence of non-technical skills assessment instruments in simulated anaesthesia crisis management. Anaesth Intensive Care. 2017 Jul;45(4):469-475. doi: 10.1177/0310057X1704500410. PMID 28673217
- [Background] Botha E, Gwin T, Purpora C. The effectiveness of mindfulness based programs in reducing stress experienced by nurses in adult hospital settings: a systematic review of quantitative evidence protocol. JBI Database System Rev Implement Rep. 2015 Oct;13(10):21-9. doi: 10.11124/jbisrir-2015-2380. PMID 26571279
- [Background] Greeson JM, Toohey MJ, Pearce MJ. An adapted, four-week mind-body skills group for medical students: reducing stress, increasing mindfulness, and enhancing self-care. Explore (NY). 2015 May-Jun;11(3):186-92. doi: 10.1016/j.explore.2015.02.003. Epub 2015 Feb 16. PMID 25792145
- [Background] Kim J, Neilipovitz D, Cardinal P, Chiu M. A comparison of global rating scale and checklist scores in the validation of an evaluation tool to assess performance in the resuscitation of critically ill patients during simulated emergencies (abbreviated as "CRM simulator study IB"). Simul Healthc. 2009 Spring;4(1):6-16. doi: 10.1097/SIH.0b013e3181880472. PMID 19212245
- [Derived] Chmielewski J, Los K, Waszkiewicz N, Luczynski W. Mindfulness Is Related to the Situational Awareness of Medical Students Confronted with Life-Threatening Emergency Situations. J Clin Med. 2021 May 2;10(9):1955. doi: 10.3390/jcm10091955. PMID 34063194
- [Derived] Los K, Chmielewski J, Cebula G, Bielecki T, Torres K, Luczynski W. Relationship between mindfulness, stress, and performance in medical students in pediatric emergency simulations. GMS J Med Educ. 2021 Apr 15;38(4):Doc78. doi: 10.3205/zma001474. eCollection 2021. PMID 34056067